CLINICAL TRIAL: NCT00111163
Title: Efficacy and Safety of Pediatric Immunization-linked Preventive Intermittent Treatment With Antimalarials in Decreasing Anemia and Malaria Morbidity in Rural Western Kenya
Brief Title: Intermittent Preventive Treatment With Antimalarials in Kenyan Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCID-3606; SSC 701
Record Dates: First submitted 2005-05-17; First posted 2005-05-18 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Malaria; Anemia
Keywords: malaria; anemia; Plasmodium falciparum; infants; prevention; safety; efficacy; antimalarials
MeSH Terms: conditions — Malaria; Anemia; Malaria, Falciparum | interventions — fanasil, pyrimethamine drug combination; Artesunate; Amodiaquine; chloroguanil, dapsone drug combination

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine with artesunate
Drug: amodiaquine with artesunate
Drug: chlorproguanil-dapsone

SUMMARY:
The purpose of the study is to see whether antimalarial drugs administered at the time of routine infant vaccinations prevents malaria and anemia in the first year of life.

DETAILED DESCRIPTION:
Approximately three quarters of preschool children in eastern Africa suffer from anemia, defined as a hemoglobin (Hb) concentration below 11 g/dL. For children < 5 years of age, the overall incidence of severe malarial anemia (Hb < 5 g/dl) is estimated at 15-60 cases per 1,000 children per year. Other studies have confirmed that the burden of malaria-related anemia falls primarily on infants and young children. In 2000, Schellenberg and colleagues, working in an area of Tanzania with a low to moderate level of Plasmodium falciparum transmission and a low level of sulfadoxine-pyrimethamine (SP) resistance, demonstrated that by linking intermittent prophylaxis to routine immunization visits through the national Expanded Program on Immunization (EPI), SP could be administered to children at 2,3, and 9 months of age, resulting in a 59% reduction in rates of clinical malaria and a 50% reduction in the rate of severe anemia (Hb<8 g/dl) compared to those receiving placebo. This randomized, double blind, placebo-controlled trial is being conducted to estimate the efficacy of Intermittent Preventive Treatment for Infants (IPTi) with SP + three doses of artesunate (AS) (SP/AS3) given in combination with iron supplementation from 2-6 months of age at routine EPI visits on the prevention of clinical malaria, moderate anemia, and severe anemia in the first 18 months of life in an area with intense malaria transmission and near universal ownership of insecticide treated nets (ITNs). The primary objective is to compare the efficacy of iron supplementation and IPTi with one of 3 antimalarial regimens (SP/AS3, chlorproguanil-dapsone (Lapdap), or AQ/AS3) given at routine EPI visits with iron supplementation alone (+ placebo) on the prevention of clinical malaria in the first year of life. Specific secondary objectives are: 1) Compare the efficacy of iron supplementation plus IPTi with one of 3 antimalarial regimens (SP/AS3, Lapdap [chlorproguanil-dapsone], or AQ/AS3) given at routine EPI visits with iron supplementation alone (+ placebo) on the prevention of moderate and severe anemia in the first year of life; 2) Assess the impact of IPTi with the aforementioned regimens on serologic responses to EPI vaccines (Polio, Diphtheria, Tetanus, Pertussis, Hepatitis B, Hemophilus Influenzae type B, and Measles; 3) Assess the impact of IPTi with the aforementioned regimens (particularly SP/AS3) on the nasal carriage rates of Haemophilus influenza type b; and 4) Compare the efficacy of iron supplementation and IPTi with one of 3 antimalarial regimens (SP/AS3, Lapdap [chlorproguanil-dapsone], or AQ/AS3) given at routine EPI visits with iron supplementation alone (+ placebo) on the prevention of all-cause hospitalization in the first year of life. This trial will generate important public health information on the efficacy of IPTi in preventing anemia and clinical malaria among infants in an area with intense malaria transmission and ongoing prevention efforts through the use of insecticide treated nets. This trial will contribute towards understanding IPTi's mechanism of action (i.e. through intermittent clearance of parasites vs. a chemoprophylactic effect afforded through the use of an antimalarial with a long half-life). The information gained will be useful to determine the safety of IPTi, and to decide what sort of antimalarials are appropriate for IPTi, and ultimately will help to direct child survival and malaria control policy in African countries. If alternative drug regimes to SP prove effective, that information will be valuable to policymakers as levels of P. falciparum resistance to SP rise with increased usage in east Africa.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for Pentavalent 1 immunization
* Age 5 weeks to 16 weeks
* Parent or guardian currently resident in study catchment area
* Parent or guardian has given permission for their child to participate

Exclusion Criteria:

* Known allergy to any of the study drugs
* Current Cotrimoxazole prophylaxis
* Concomitant disease requiring hospitalization or transfusion
* Plans to be away from the study area for more than 6 months during the next year

Ages: 5 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1516
Dates: Start 2004-03; Primary Completion 2006-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Clinical malaria in the first year of life

SECONDARY OUTCOMES:
Moderate and severe anemia in the first year of life
Serologic responses to Expanded Program on Immunization (EPI) vaccines (Polio, Diphtheria, Tetanus, Pertussis, Hepatitis B, Hemophilus Influenzae type B, and Measles)
Nasal carriage rates of Haemophilus influenza type b
All cause hospitalization in the first year of life

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Newman, MD, MPH, Principal Investigator — U.S. Centers for Disease Control and Prevention; Laurence Slutsker, MD, MPH, Principal Investigator — U.S. Centers for Disease Control and Prevention
Locations (1):
- Lwak, Abidha, Ongielo and Saradidi clinics, Asembo (Rarieda Division), Nyanza Province, Kenya

REFERENCES:
- [Background] Schellenberg D, Menendez C, Kahigwa E, Aponte J, Vidal J, Tanner M, Mshinda H, Alonso P. Intermittent treatment for malaria and anaemia control at time of routine vaccinations in Tanzanian infants: a randomised, placebo-controlled trial. Lancet. 2001 May 12;357(9267):1471-7. doi: 10.1016/S0140-6736(00)04643-2. PMID 11377597
- [Background] Massaga JJ, Kitua AY, Lemnge MM, Akida JA, Malle LN, Ronn AM, Theander TG, Bygbjerg IC. Effect of intermittent treatment with amodiaquine on anaemia and malarial fevers in infants in Tanzania: a randomised placebo-controlled trial. Lancet. 2003 May 31;361(9372):1853-60. doi: 10.1016/s0140-6736(03)13504-0. PMID 12788572
- [Derived] Odhiambo FO, Hamel MJ, Williamson J, Lindblade K, ter Kuile FO, Peterson E, Otieno P, Kariuki S, Vulule J, Slutsker L, Newman RD. Intermittent preventive treatment in infants for the prevention of malaria in rural Western kenya: a randomized, double-blind placebo-controlled trial. PLoS One. 2010 Apr 2;5(4):e10016. doi: 10.1371/journal.pone.0010016. PMID 20368815
- See also: Website for the Intermittent Preventive Treatments in Infants (IPTi) Consortium, assisting in development of comprehensive research and implementation agenda — http://www.ipti-malaria.org/